CLINICAL TRIAL: NCT00705471
Title: Infliximab Use in Fistulizing Crohn's Disease: Impact on Health Care Resources
Brief Title: Impact of Infliximab in Fistulizing Crohn's Disease on Health Care Resources (Study P04204)(TERMINATED)
Status: Terminated | Type: Observational
Why Stopped: Study stopped prematurely due to enrolment challenges.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P04204
Record Dates: First submitted 2008-06-23; First posted 2008-06-26 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab: Because of the difficulty of finding subjects with exactly the same disease severity, information will be recorded for the time period for up to three years before and for one year after their initial infliximab infusion for comparison of health care costs and utilization prior to infliximab and post infliximab use.
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — None available in the protocol. This was a chart review study, therefore no Infliximab provided during the study.
  Other Names: Remicade; SCH 215596

SUMMARY:
A multi-centre retrospective review of fistulizing Crohn's disease (CD) patient charts will capture data to measure health care resource utilization associated with the use of Infliximab for treatment of CD. Three health science centres/hospitals from Ontario are targeted to participate in the study, each site is expected to provide 30-40 patient charts with a target of 108 charts total.

DETAILED DESCRIPTION:
This study population was chosen from a non-probability sample.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with infliximab for fistulizing CD.
* Administration of at least one infliximab infusion >=12 months before the chart review.
* 18 years of age or over (men and women).

Exclusion Criteria:

* Subjects not followed for a full year after their first infusion of infliximab.
* Subjects not followed for a full year prior to their first infusion of infliximab.
* Subjects who had participated in clinical studies during the data collection timeframe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The charts of subjects with fistulizing CD to be recorded for the time period for up to three years before and for one year after their initial infliximab infusion for comparison of health care costs and utilization prior to infliximab and post infliximab use.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2005-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To quantify the impact of infliximab therapy on the Canadian healthcare resource utilization as expressed as incidence per year. | 1 year

SECONDARY OUTCOMES:
To quantify the impact of infliximab therapy on healthcare resource utilization as expressed in Canadian dollars. | 1 year